

## Project manager:

Dr. Barbara Vona Institute for Auditory Neuroscience Robert-Koch-Str. 40 37075 Göttingen, Germany Tel: (+49) 551-38-51337 Email: barbara.vona@med.uni-goettingen.de

### **Institute for Auditory Neuroscience**

Director: Prof. Dr. Tobias Moser Robert-Koch-Str. 40, 37075 Göttingen, Germany

### Department of Otolaryngology

Prof. Dr. med. Nicola Strenzke Robert-Koch-Str. 40, 37075 Göttingen, Germany

#### **Institute of Human Genetics**

Director: Prof. Dr. med. Bernd Wollnik Heinrich-Düker-Weg 12, 37073 Göttingen, Germany

ClinicalTrials.gov Identifier: NCT06680934

May 16<sup>th</sup>, 2025

# CABP2 Registry

# What is the CABP2 Registry?

The *CABP2* Registry collects clinical information (various hearing tests and medical information) as well as genetic (Calcium-binding protein 2, *CABP2*) mutation details for research and therapy development. Through consent and participation, the *CABP2* Registry aims to advance scientific knowledge by connecting (pseudonymized) patient data with scientists at the Institute for Auditory Neuroscience at University Medical Center Goettingen who have shown decades-long interest in understanding the mechanisms of several forms of hereditary hearing impairment, among which includes *CABP2*.

In a collaboration between the Institute for Auditory Neuroscience and the Institute of Human Genetics at University Medical Center Goettingen, we have initiated a study wherein we aim to collect and evaluate the clinical and genetic findings of individuals with mutations in the *CABP2* gene. This will allow us to better understand the relationship between mutations and hearing loss and to improve patient care as new therapies are optimized. To support this goal, we have established a patient registry for voluntary participation and sharing of clinical and genetic information in questionnaire form.

This registry study was approved by the Ethics Committee of the University Medical Center Goettingen (Approval: 17/8/22; Study Center ID: 2023-02528).

# Who can participate in the CABP2 Registry?

The *CABP*2 Registry is open to the global *CABP*2 community that includes parents and legal guardians, as well as individuals who have been diagnosed with hearing impairment due to *CABP*2 mutations.

## Where can participants find out more information?

We invite prospective participants to review detailed study information and submit consent (<a href="http://www.auditory-neuroscience.uni-goettingen.de/cabp2">http://www.auditory-neuroscience.uni-goettingen.de/cabp2</a> registry en.html). This also includes information about the processing of personal data.

### Who can participants contact for more information?

If you have questions or would like further clarification about the procedure, please contact the study manager, Dr. Barbara Vona, via email: barbara.vona@med.uni-goettingen.de.